CLINICAL TRIAL: NCT03945227
Title: A Phase II Clinical Trial for Evaluating Efficacy and Safety of PDR001 in Concurrent Plus Consolidation Versus Consolidation Only in Addition to Standard Chemoradiotherapy in Unresectable Stage III NSCLC Patients (PASTURE)
Brief Title: Clinical Trial for Evaluating Efficacy and Safety of PDR001 in Concurrent Plus Consolidation Versus Consolidation Only in Addition to Standard Chemoradiotherapy in Unresectable Stage III NSCLC Patients (PASTURE)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the delay in the study shceduled, due to the start of competitive study and the approval of Durvalumab from the Ministry of Food and Drug Safety, it was judged that it was difficult to enroll subjects.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-1171
Record Dates: First submitted 2019-04-24; First posted 2019-05-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stage III NSCLC
Keywords: Non small cell lung cancer; Unresectable stage III NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (consolidation only arm) (Placebo Comparator): Arm A (consolidation only arm) will be treated with standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001 regimen. --For concurrent chemoradiation therapy, chemotherapeutic agents will follow the one of the two regimens of standard of care Paclitaxel 45 mg/m2 at D1, D8, D15, D22, D29, and D36, IV infusion; Carboplatin AUC 2 at D1, D8, D15, D22, D29, and D36, IV infusion Etoposide 50 mg/m2 D1-5, D29-33,IV infusion; Cisplatin 50 mg/m2 D1, D8, D29, and D36; IV infusion - Concurrent radiation therapy (generally, 60 Gy/30 Fx ±10%) - Consolidation therapy: after 2 weeks after completion of radiation therapy (± 7 days), PDR001 400 mg every 4 weeks, until disease progression or an unacceptable adverse event, maximum 12 months.
  Interventions: Drug: standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001
- Arm B (concurrent arm) (Experimental): Arm B (concurrent arm) will be treated with PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001 regimen. --For concurrent chemoradiation therapy, chemotherapeutic agents will follow one of the two regimens of standard of care Paclitaxel 45 mg/m2 at D1, D8, D15, D22, D29, and D36, IV infusion; Carboplatin AUC 2 at D1, D8, D15, D22, D29, and D36, IV infusion Etoposide 50 mg/m2 D1-5, D29-33,IV infusion; Cisplatin 50 mg/m2 days 1,8,29, and 36; IV infusion - Concurrent PDR001 400mg at D1, D29 - Concurrent radiation therapy (generally, 60 Gy/30 Fx ±10%) - Consolidation therapy: after 4 weeks after last dose of PDR001, PDR001 400 mg every 4 weeks, until disease progression or an unacceptable adverse event, maximum 12 months.
  Interventions: Drug: PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001

INTERVENTIONS:
Drug: standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001 — drug: standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001 Arm A (consolidation only arm) will be treated with standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001 regimen. --For concurrent chemoradiation therapy, chemotherapeutic agents will follow the one of the two regimens of standard of care Paclitaxel 45 mg/m2 at D1, D8, D15, D22, D29, and D36, IV infusion; Carboplatin AUC 2 at D1, D8, D15, D22, D29, and D36, IV infusion Etoposide 50 mg/m2 D1-5, D29-33,IV infusion; Cisplatin 50 mg/m2 D1, D8, D29, and D36; IV infusion - Concurrent radiation therapy (generally, 60 Gy/30 Fx ±10%) - Consolidation therapy: after 2 weeks after completion of radiation therapy (± 7 days), PDR001 400 mg every 4 weeks, until disease progression or an unacceptable adverse event, maximum 12 months.
  Arms: Arm A (consolidation only arm)
Drug: PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001 — drug:PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001 Arm B (concurrent arm) will be treated with PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001 regimen. -For concurrent chemoradiation therapy, chemotherapeutic agents will follow one of the two regimens of standard of care Paclitaxel 45 mg/m2 at D1, D8, D15, D22, D29, and D36, IV infusion; Carboplatin AUC 2 at D1, D8, D15, D22, D29, and D36, IV infusion Etoposide 50 mg/m2 D1-5, D29-33,IV infusion; Cisplatin 50 mg/m2 days 1,8,29, and 36; IV infusion - Concurrent PDR001 400mg at D1, D29 - Concurrent radiation therapy (generally, 60 Gy/30 Fx ±10%) - Consolidation therapy: after 4 weeks after last dose of PDR001, PDR001 400 mg every 4 weeks, until disease progression or an unacceptable adverse event, maximum 12 months.
  Arms: Arm B (concurrent arm)

SUMMARY:
This is a multi-center, open-label, randomized Phase 2 trial evaluating PDR001 in two arms for concurrent chemoradiation and consolidation in the treatment-naïve patients with locally advanced, unresectable stage III NSCLC. Patients will be randomized in a 1:1 ratio (arm A and arm B):

* Arm A (consolidation only arm) will be treated with standard platinum-based concurrent chemoradiotherapy, followed by consolidation with PDR001 regimen.
* Arm B (concurrent arm) will be treated with PDR001 concurrent with standard platinum-based chemoradiation, followed by consolidation with PDR001 regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cytologically or histologically proven, locally advanced, treatment-naïve, unresectable, both squamous and non-squamous stage III NSCLC* (According to AJCC TNM staging 8th edition, IIIB and IIIC diseases are eligible; Inoperable stage IIIA disease without any exclusion criteria is also eligible)
2. Patients with targetable mutations such as EGFR, ALK and ROS1 are also eligible
3. Measurable disease based on RECIST 1.1 as determined by the site.
4. Men and women ≥ 20 years of age
5. A performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) performance Status
6. Adequate hematologic, renal, and hepatic function as follows:

   * Absolute Neutrophil Count (ANC), > 1,000/mm3
   * Platelets > 100,000/mm3
   * Hemoglobin > 9.0 g/dL
   * Serum creatinine < 1.5 × upper normal limit (ULN) OR creatinine clearance > 45 mL/min/1.73m2
   * AST and/or ALT < 2.5 × the ULN
   * Bilirubin < 1.5 × the ULN
7. 12-Lead electrocardiogram (ECG) shows QTc interval ≤470 msec and without history of Torsades de Pointes or other symptomatic QTc abnormality
8. Written (signed) Informed Consent to participate in the study

Exclusion Criteria:

1. Prior exposure to any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associate antigen-4 (CTLA-4) antibody
2. Active or prior autoimmune disease or history of immunodeficiency
3. Current or prior use of immunosuppressive agents within 28 days before the first dose of investigational drugs, with the exception of intranasal, inhaled, or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
4. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GMCSF, M-CSF), thrombopoietin mimetics or erythroid stimulating agents ≤ 2 weeks prior start of study treatment. If erythroid stimulating agents were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained
5. Experience of solid organ transplant
6. Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
7. Evidence of uncontrolled illness such as symptomatic congestive heart failure, uncontrolled hypertension or unstable angina pectoris.
8. Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis)
9. Active infection of lung, including pulmonary tuberculosis, pneumonia
10. Has a history of interstitial lung disease (ILD) or a history of pneumonitis that has required oral or IV steroids.
11. Pregnant female subject (Female subjects must have a negative urine or serum pregnancy test at screening if of childbearing potential, or be of non-child bearing potential.)
12. Lactating female subject
13. Prior malignancy, with the exception of basal cell/ squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 3 years since initiation of that therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival (PFS) | Repeated tumor imaging will be performed every 8 weeks from randomization until the date of disease progression or up to 18 months. And Tumor Imaging Change will assessed by RECIST 1.1
  To compare the progression free survival (PFS) in concurrent plus consolidation PDR001 vs. consolidation PDR001 only in addition to standard platinum-based concurrent chemoradiation, in the patients with locally advanced, unresectable stage III NSCLC.

SECONDARY OUTCOMES:
To evaluate antitumor efficacy of PDR001: OS | Repeated tumor imaging will be performed every 8 weeks from randomization until the date of disease progression or up to 18 months. And Tumor Imaging Change will assessed by RECIST 1.1
  To evaluate the overall survival (OS) of PDR001 as concurrent plus consolidation versus consolidation only treatment in addition to platinum-based concurrent chemoradiation, in the patients with locally advanced, unresectable stage III NSCLC.
To evaluate antitumor efficacy of PDR001: ORR | Repeated tumor imaging will be performed every 8 weeks from randomization until the date of disease progression or up to 18 months. And Tumor Imaging Change will assessed by RECIST 1.1
  To compare objective response rate (ORR; evaluated by RECIST) of the patients who received platinum-based concurrent chemoradiation with or without concurrent PDR001.
Incidence of Treatment-Emergent Adverse Events[Safety and Tolerability) | Repeated tumor imaging will be performed every 8 weeks from randomization until the date of disease progression or up to 18 months. And Tumor Imaging Change will assessed by RECIST 1.1
  To evaluate the safety and tolerability profile of PDR001 as concurrent plus consolidation versus consolidation only treatment in addition to platinum-based concurrent chemoradiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Yonsei University College of Medicine, Seoul, South Korea